CLINICAL TRIAL: NCT03504150
Title: Comparative Effectiveness of Two Self-guided Web-based Interventions for Youth and Young Adults With Migraine
Brief Title: Testing myWHI: Online Self-help Programs for Headaches
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IWK Health Centre (Other)
Collaborators: Nova Scotia Health Research Foundation (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Anna Huguet, Principal investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1022640
Record Dates: First submitted 2018-04-05; First posted 2018-04-20 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPHERE (Experimental): It is an online self-guided comprehensive cognitive-behavioural therapy program that offers a headache diary, learning modules that teach a variety of cognitive and behavioural skills to cope better with their headaches, and a discussion forum where users may interact.
  Interventions: Behavioral: SPHERE
- PRISM (Experimental): It is an online self-guided brief cognitive-behavioural therapy program that offers a headache diary and helps users discover their headache triggers and non-triggers. Then the program provides the users with a few personalized recommendations to help them to cope with their triggers.
  Interventions: Behavioral: PRISM
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: SPHERE — Comprehensive Internet-based CBT program with no human support
  Arms: SPHERE
Behavioral: PRISM — Brief Internet-based CBT program with no human support
  Arms: PRISM

SUMMARY:
This randomized controlled trial will compare the effectiveness of two online self-guided programs for youth and young adults with migraine against usual care.

ELIGIBILITY:
Inclusion criteria:

* aged 14-40 years
* fluent in the English language (i.e., speaking, reading and writing);
* for 14-17 year olds: suffer from headaches for a minimum of three months
* for 18-40 year olds: suffer from headaches for a minimum of one year
* suffer from migraine headaches as indicated with a score of 2 and above on the ID Migraine
* have a Smartphone as PRISM has been designed to be accessed from a Smartphone and SPHERE encompasses the myWHI diary which has also been designed to be used from a Smartphone
* use the Smartphone for activities other than texting and calling (e.g., email, Facebook) as the programs are designed for migraineurs who are familiar with using Smartphones and use them in their daily life
* have daily Internet access from their Smartphone, because running the programs require an Internet connection
* minimum of four headache days during 4 weeks that they are asked to use an electronic headache diary

Exclusion criteria:

* health care professional has not ruled out any underlying medical condition related to their headaches (e.g., head trauma, meningitis)
* are pregnant, planning to get pregnant (in the next 4 to 6 months), or breastfeeding, as hormonal changes are known to exert potent influences on migraine headaches
* have an impairment which compromises their ability to give informed consent
* having been diagnosed with psychosis and/or schizophrenia, because a past or current diagnosis may likely interfere with the participants ability to fully participate in the study
* have participated in our recent three-armed pilot RCT (i.e., any participant who consented and was randomized)
* they complete less than 50% of daily entries (i.e., less than 14 daily entries) in an electronic headache dairy when they asked to use it for 4 weeks
* More than 15 headache days during the 4 weeks that they are asked to use an electronic headache diary

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants will be asked:
  Are you: Male, Female, or I do not want to answer this question
Enrollment: 424 (Estimated)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Clinically significant improvement (50% reduction or greater) in number of headache days in a 4-week period from baseline to 4-months post-randomization | At baseline and at 4-months post-randomization
  An electronic headache diary will be asked to be used for 4 weeks. Each day participants will be asked to record whether or not they have experienced a headache.

SECONDARY OUTCOMES:
Statistically significant improvement in peak headache severity in a 4-week period from baseline to 4-months post-randomization | At baseline and at 4-months post-randomization
  An electronic headache diary will be asked to be used for 4 weeks. On days that participants report a headache(s) in the diary, they will be asked to rate highest headache intensity for the day using the 11-point Numerical Rating Scale (NRS-11). The peak headache severity will be calculated in two different ways: (1) the average of the highest headache intensity per week over the 4-week period, and (2) the number of days that participants have reported a headache episode with a NRS-11 of 8 or higher over the 4-week period.
Statistically significant improvement in headache-related functional impairment from baseline to 4-months post-randomization | At baseline and at 4-months post-randomization
  We will measure impairment with either the Migraine Disability Assessment Scale -Pediatric version (PedMIDAS) for ages 14-18 years or the Migraine Disability Assessment Scale (MIDAS) for ages 19-40 years. MIDAS and PedMIDAS measure headache-related functional impairment. We will use the total score, which is the sum of answers across the 6 items for PedMIDAS and the sum of answers across the 5 items for MIDAS. A higher score indicating greater impairment.
Statistically significant improvement in depressive symptomatology from baseline to 4-months post-randomization. | At baseline and at 4-months post-randomization
  The Centre for Epidemiological Studies - Depression Scale (CES-D) will be used to measure depressive symptomatology. Responses will be summed to provide a total score that can range from 0 to 60; with higher scores indicating the presence of more symptoms and higher frequency.
Level of acceptability to the treatments (i.e., PRISM and SPHERE) | At 4-months post-randomization
  The 8-item Client Satisfaction Questionnaire (CSQ-8) will be used to measure level of acceptability to the treatments. The total score will be used. The total score is the sum of item responses and ranges from 8 to 32, with higher scores indicating higher levels of satisfaction.
Level of acceptability to the treatments (i.e., PRISM and SPHERE) | At 4-months post-randomization
  The single-item Patients' Global Impression of Change (PGIC) Scale will be used to measure level of acceptability to the treatments. The PGIC is 7-point categorical scale ("very much improved" to "very much worse") to report the perceived improvement with an intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Huguet, PhD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No